CLINICAL TRIAL: NCT06711887
Title: An Open-label Extension Study to Assess the Efficacy and Safety of Ianalumab With or Without Study Treatment Withdrawal in Adult Participants With Lupus Nephritis Who Have Completed Study Treatment in the CVAY736K12301 Core Study (SIRIUS-LN Extension)
Brief Title: Phase III Extension Study of Efficacy and Safety of Ianalumab With or Without Study Treatment Withdrawal in Participants With Lupus Nephritis (SIRIUS-LN Extension)
Acronym: SIRIUS-LN ext
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAY736K12301E1
Expanded Access: NCT07244289 (Available)
Record Dates: First submitted 2024-11-11; First posted 2024-12-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis (LN); B cell depletion; ianalumab; VAY736
MeSH Terms: conditions — Lupus Nephritis | interventions — ianalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Study Treatment Withdrawal (cohort 1) (No Intervention): (Cohort 1): Study Treatment-Withdrawal group. Participants who received blinded study treatment in the core study and achieve CRR or PRR at Week 140 in the core study will enter the extension study and discontinue study treatment while maintaining standard of care (SoC) medication, as required. If renal flare criteria are met, participants will be eligible to receive open-label ianalumab.
- Open-Label Ianalumab (cohort 2) (Experimental): (Cohort 2): Open-Label Ianalumab group: Participants who received blinded study treatment throughout the core study and did not achieve CRR or PRR at Week 140 of the core study, or who had switched to open-label ianalumab during the core study, will be eligible or will continue to receive open-label ianalumab in the extension study.
  Interventions: Drug: Ianalumab

INTERVENTIONS:
Drug: Ianalumab — Ianalumab (VAY736) is a human monoclonal antibody (mAb) of the IgG1/κ-class, directed against B cells and binding to BAFF receptor (BAFF-R).
  Other Names: VAY736
  Arms: Open-Label Ianalumab (cohort 2)

SUMMARY:
The purpose of this 2-year extension study is the evaluation of the efficacy and safety

1. after study treatment withdrawal in patients with lupus nephritis (LN) who achieved response (complete renal response [CRR] or partial renal response [PRR]) on double-blind treatment at the end of the SIRIUS-LN core study, and
2. of open-label ianalumab 300 mg treatment in patients who, at the end of the SIRIUS-LN core study, were either already receiving ianalumab open-label treatment or did not meet CRR/PRR criteria on double-blind treatment at the end of the SIRIUS-LN core study.

DETAILED DESCRIPTION:
The SIRIUS-LN extension study is a 2-year open-label extension study for participants who have completed the treatment periods (blinded Treatment Period-1 and blinded Treatment Period-2) of the SIRIUS-LN core study on double-blind or open-label study treatment.

Investigators will use their clinical judgment to decide if it is beneficial for participants to continue with the extension study. In this extension study participants who achieve CRR or PRR status at Week 140 will be withdrawn from study treatment and will maintain the SoC medication as required. These 2 additional years in the extension study will allow to measure sustained remission, flares and safety off-study treatment. However, in the event of renal flares during the extension study, these participants who withdraw study treatment will have the option to receive open-label ianalumab.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the extension study.
2. Participants must have participated in the SIRIUS-LN core study and must have completed the entire treatment up to Week 144 on double-blind or open label study treatment.

Exclusion Criteria:

1. Use of prohibited therapies
2. Pregnant or nursing (lactating) women.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2030-07-16 (Estimated); Study Completion 2032-07-16 (Estimated)

PRIMARY OUTCOMES:
For cohort 1: Incidence of renal flare, escalation of immunosuppressive medication, or death | Between Week 144E1 and Week 248
  Cohort 1: To estimate the incidence of renal flare, escalation of immunosuppressive medication, or death following study treatment withdrawal in participants who completed the SIRIUS-LN core study on double-blind treatment and achieved CRR or PRR at Week 140 of the core study
Cohort 2: Number of participants with Treatment Emergent Adverse Events (TEAE) as assessed by CTAE v4.0 | From the start of treatment in the SIRIUS-LN core study to EOS (up to week 352) of the extension study
  Cohort 2: To assess the safety and tolerability of ianalumab for participants who, at the end of the SIRIUS-LN core study, were either already receiving ianalumab open-label treatment or did not meet CRR/PRR criteria on double-blind treatment at the end of the SIRIUS-LN core study
Cohort 2: Number of participants with Serious Adverse Events (SAE) as assessed by CTCAE v4.0 | From the start of treatment in the SIRIUS-LN core study to EOS (up to week 352) of the extension study
  Cohort 2: Incidence of SAEs, from the start of treatment in the SIRIUS-LN core study to EOS (up to week 352) of the extension study
Cohort 2: Number of participants with clinically significant abnormal vital signs | From the start of treatment in the SIRIUS-LN core study to EOS (up to week 352) of the extension study
  Cohort 2: Analysis of the vital sign measurements using summary statistics for the change from baseline for each post-baseline visit will be performed
Cohort 2: Number of participants with clinically significant laboratory evaluations. | From the start of treatment in the SIRIUS-LN core study to EOS (up to week 352) of the extension study
  Cohort 2: The summary of laboratory evaluations will be presented for two groups of laboratory tests (hematology and serum chemistry). Descriptive summary statistics for the change from baseline to each study visit will be presented. These descriptive summaries will be presented by test group, laboratory test and treatment group.

SECONDARY OUTCOMES:
Cohort 1: Number of participants with Treatment Emergent Adverse Events (TEAE) as assessed by CTCAE v4.0 | From the start of treatment in the SIRIUS-LN core study up to EOS (week 248) of the extension study
  To assess the safety and tolerability of ianalumab in Cohort 1
Cohort 2: Incidence and titer of anti-ianalumab antibodies in serum (ADA assay) | from Week 144E1 up to Week 248
  To assess immunogenicity to ianalumab in Cohort 2
Cohort 2: Ianalumab concentration in serum using a validated ELISA | from Week 144E1 up to Week 248
  To assess pharmacokinetics of ianalumab in Cohort 2
Cohort 1: Number of participants with Serious Adverse Events (SAE) as assessed by CTAE v4.0 | From the start of treatment in the SIRIUS-LN core study up to EOS (week 248) of the extension study
  To assess the safety and tolerability of ianalumab in Cohort 1
Cohort 1: Number of participants with clinically significant abnormal vital signs | From the start of treatment in the SIRIUS-LN core study up to EOS (week 248) of the extension study
  To assess the safety and tolerability of ianalumab in Cohort 1
Cohort 1: Number of participants with clinically significant abnormal laboratory evaluations | From the start of treatment in the SIRIUS-LN core study up to EOS (week 248) of the extension study
  To assess the safety and tolerability of ianalumab in Cohort 1

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (17):
- China (5):
  - Novartis Investigative Site, Liuchow, Guangxi
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Binzhou, Shandong
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
- Novartis Investigative Site, Barranquilla, Atlántico, Colombia
- Novartis Investigative Site, Budapest, Hungary
- Mexico (3):
  - Novartis Investigative Site, León, Guanajuato
  - Novartis Investigative Site, Oaxaca City
  - Novartis Investigative Site, Querétaro
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Taichung, Taiwan
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Ahmad SB, Jefferson JA. Targeting B Cells and Plasma Cells in Glomerular Disease. J Am Soc Nephrol. 2025 Jun 4;36(9):1844-1857. doi: 10.1681/ASN.0000000772. PMID 40465397